CLINICAL TRIAL: NCT05576285
Title: Retinal Imaging Study of Children That Might be at Risk of Having Retinal Hemorrhages
Acronym: RISC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Kerstin Hellgren, Associate professor, Region Stockholm
Other Study IDs: Dnr 2022-00506-01
Record Dates: First submitted 2022-09-29; First posted 2022-10-12 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Retinal Hemorrhage, Bilateral; Retinal Hemorrhage, Left Eye; Retinal Hemorrhage, Right Eye
Keywords: retinal hemorrhage
MeSH Terms: conditions — Retinal Hemorrhage | interventions — Ophthalmoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Accelerating head growth in infancy: Infants <=18 months of age referred to head ultrasound because of accelerating head growth
  Interventions: Diagnostic Test: ophthalmoscopy and fundus photography through dilated pupills
- Children at ICU with neurological symptoms that require brain MRI or CT: Children < 15 years of age who are cared for at ICU becaus of neurological symptoms that require brain MRI or CT scans
  Interventions: Diagnostic Test: ophthalmoscopy and fundus photography through dilated pupills
- Children entering the emergency department with the need of acute brain CT: Children < 2 years of age that enter the emergency department because of brainthreatening conditions that require acute brain CT scans
  Interventions: Diagnostic Test: ophthalmoscopy and fundus photography through dilated pupills

INTERVENTIONS:
Diagnostic Test: ophthalmoscopy and fundus photography through dilated pupills — ophthalmoscopy and fundus photography through dilated pupills

SUMMARY:
This is a clinical trial in which we will learn about the retinal findings in three clinical groups of children, who might be at risk of having retinal hemorrhages (RH). The aim of the study is to explore the occurrence of moderate to severe retinal hemorrhages in critically ill children, children with intracranial hemorrhages, hydrocephalus or signs of elevated intracranial pressure and in children with benign enlargement of subarachnoid spaces (BESS).

1. Are RHs associated with BESS?
2. What is the prevalence, distribution and extent of RHs in critically ill children?
3. What is the prevalence, distribution and extent of RHs in children with traumatic brain injury?
4. Does the prevalence, distribution and extent of RHs differ in children with witnessed traumatic brain injury from children with traumatic brain injury of unknown origin?
5. To what extent do the causes of RHs affect visual acuity, initially and during recovery? A retinal ophthalmoscopy through dilated pupils will be conducted and a fundus photograph will be taken by a handheld, non-touch camera.

DETAILED DESCRIPTION:
The prospective study will take place at university hospitals in three Swedish regions, Stockholm, Skåne and Västra Götaland. The data collection from the three regions will proceed in parallel over a three-year period. An estimated number of children will be 400-500 per year. The study children will be consecutively referred to the pediatric ophthalmology units, where the ophthalmological examinations will take place. Bedside examinations will be performed when indicated at the pediatric intensive care units. Retinal fundus examination will be performed according to clinical standards following administration of pupil dilating eye drops in each eye. Visual function will be evaluated if ophthalmic abnormalities are detected.

Prospective observational study Group 1: All infants ≤ 18 months of age, who undergo neuroradiological examinations of the brain on the indication increased head circumference.

Group 2: All critically ill children < 15 years of age, cared for at the hospitals, with neurological symptoms, that require neuroradiological examination of the brain.

Group 3: All children ≤ 2 years of age, who undergo emergency neuroradiological examinations of the head at the hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤ 18 months of age, who undergo neuroradiological examinations of the brain on the indication increased head circumference
* Children < 15 years of age, cared for at the ICU, with neurological symptoms, that require neuroradiological examination of the brain
* Children < 5 years of age, who undergo emergency neuroradiological examinations of the head at the hospitals

Exclusion Criteria

- Infants with intraventricular hemorrhages due to prematurity, in the absence of increased head circumference

Ages: 4 Weeks to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Residents in the Stockholm region, the Skåne region and the Västra Götaland region
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with retinal hemorrhages | 20 minutes
  Ophthalmoloscopy findings registered in protocol and fundus photographs
Number and distribution of retinal hemorrhages in eyes | 20 minutes
  Ophthalmoloscopy findings registered in protocol and fundus photographs

SECONDARY OUTCOMES:
Visual function | 10 minutes
  Following and fixating LH face
Eye movements | 10 minutes
  Following and fixating LH face

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin M Hellgren, MD, PhD, Principal Investigator — Region Stockholm
Locations (1):
- Kerstin Margareta Hellgren, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No